CLINICAL TRIAL: NCT02919319
Title: Double-blind, Placebo-controlled, Randomized, Single Ascending Dose Study to Investigate the Tolerability, Safety, Pharmacokinetics, Pharmacodynamics, Absolute Bioavailability, Mass Balance, and Metabolism of ACT-541468 in Healthy Male Subjects
Brief Title: A Single Ascending Dose Study of ACT-541468 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: AC-078-101; 2014-003129-16 (EudraCT Number)
Record Dates: First submitted 2016-09-28; First posted 2016-09-29 (Estimated); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — daridorexant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (5):
- Dose group 1 (Experimental): Six subjects received 5 mg of ACT-541468 (formulation A) as a single oral dose and two subjects received the matching placebo.
  Interventions: Drug: ACT-541468 (Formulation A); Drug: Placebo (Formulation A)
- Dose group 2 (Experimental): Three subjects received a single oral dose (25 mg) of ACT-541468 formulation A during Period 1 and a single oral dose (25 mg) of ACT-541468 formulation B during Period 2. Three other subjects Subjects received ACT-541468 formulation B during Period 1 and ACT-541468 formulation A during Period 2. Two additional subjects received the matching placebos in both treatment periods.
  Interventions: Drug: ACT-541468 (Formulation A); Drug: ACT-541468 (Formulation B); Drug: Placebo (Formulation A); Drug: Placebo (Formulation B)
- Dose group 3 (Experimental): Six subjects received 50 mg of ACT-541468 (formulation A) as a single oral dose in combination with a [14C]-ACT-541468 oral tracer for the mass balance and metabolism analyses. Two other subjects received the matching placebos.
  Interventions: Drug: ACT-541468 (Formulation A); Drug: Placebo (Formulation A); Drug: 14C-labeled ACT-541468; Drug: Placebo tracer
- Dose group 4 (Experimental): Six subjects received 100 mg of ACT-541468 (formulation A) as a single oral dose in combination with a [14C]-ACT-541468 intravenous tracer for the absolute bioavailability assessment. Two other subjects received the matching placebos.
  Interventions: Drug: ACT-541468 (Formulation A); Drug: Placebo (Formulation A); Drug: 14C-labeled ACT-541468; Drug: Placebo tracer
- Dose group 5 (Experimental): Six subjects received 200 mg of ACT-541468 (formulation A) as a single oral dose and two subjects received the matching placebo.
  Interventions: Drug: ACT-541468 (Formulation A); Drug: Placebo (Formulation A)

INTERVENTIONS:
Drug: ACT-541468 (Formulation A) — Hard gelatin capsules for oral administration formulated at strengths of 5 mg, 25 mg and 100 mg
Drug: ACT-541468 (Formulation B) — Soft gelatin capsules for oral administration formulated at the strength of 25 mg
  Arms: Dose group 2
Drug: Placebo (Formulation A) — Hard capsules matching ACT-541468 Formulation A
Drug: Placebo (Formulation B) — Soft capsules matching ACT-541468 Formulation B
  Arms: Dose group 2
Drug: 14C-labeled ACT-541468 — Tracer at a nominal dose of 250 nCi (corresponding to 2.02 µg ACT-541468) administered either orally or intravenously
  Arms: Dose group 3; Dose group 4
Drug: Placebo tracer — Sterile NaCl 0.9% was used as placebo matching the tracer for oral and i.v. administration.
  Arms: Dose group 3; Dose group 4

SUMMARY:
The main objectives of this first-into-man study were to investigate the safety, tolerability and the pharmacokinetic profile of single oral doses of ACT-541468 in healthy male adults. Pharmacodynamic effects (through a battery of Central Nervous System tests) were also assessed.

DETAILED DESCRIPTION:
The study consisted of ascending dose groups; each dose group was investigated in a new group of 8 healthy male subjects (6 on active drug and 2 on placebo). In addition, the study included a biocomparison part (dose group 2), an absolute bioavailability part (dose group 4), and a mass balance / metabolism part (dose group 3).

ELIGIBILITY:
Key inclusion Criteria:

* Signed informed consent prior to any study-mandated procedure.
* Males aged from 18 to 45 years (inclusive) at screening.
* Body mass index (BMI) between 18.0 and 30.0 kg/m2 (inclusive) at screening.
* Systolic blood pressure (SBP), diastolic blood pressure (DBP) and pulse rate (PR) between 100-145 mmHg, 50-90 mmHg and 45-90 bpm (all inclusive) at screening, respectively.
* Healthy on the basis of physical examination,electrocardiogram and laboratory tests.

Key exclusion Criteria:

* Known hypersensitivity to any excipients of the drug formulations.
* History or presence of any disease or condition or treatment, which may put the subject at risk of participation in the study or may interfere with the absorption, distribution, metabolism or excretion of the study drugs.
* History of narcolepsy or cataplexy or modified Swiss narcolepsy scale total score < 0 at screening.
* Any circumstances or conditions, which, in the opinion of the investigator, may affect the subject's full participation in the study or compliance with the protocol.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2015-05-01 (Actual); Study Completion 2015-05-01 (Actual)

PRIMARY OUTCOMES:
Number of subjects with treatment-emergent adverse events and serious adverse events | Day 8
  Collection of any adverse event at each dose level

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of ACT-541468 | From pre-dose up to 168 hours post-dose
  Cmax was directly derived from the observed plasma concentrations of ACT-541468 for each dose level
Time to reach Cmax (tmax) of ACT-541468 | From pre-dose up to 168 hours post-dose
  tmax was directly derived from the observed plasma concentrations of ACT-541468 for each dose level
Terminal half-life (t1/2) of ACT-541468 | From pre-dose up to 168 hours post-dose
  t1/2 was calculated from the terminal rate constant obtained from the plasma concentrations-time curves of ACT-541468, at each dose level
Area under the plasma concentration-time curves [AUC(0-inf)] of ACT-541468 | From pre-dose up to 168 hours post-dose
  AUC(0-inf) is the area under the plasma concentration-time curves of ACT-541468, calculated from time 0 (pre-dose) to extrapolated infinite time, at each dose level
Percentage of dose excreted in feces and urine | From pre-dose up to 168 hours post-dose
  Percentage of oral dose of 14C-labeled ACT-541468 excreted in feces (FPE), urine (UPE) and both, as determined in the dose group 3
Absolute bioavailability (F) of ACT-541468 | Up to 96 hours post-dose
  Absolute bioavailability was determined for dose group 4 and defined as the ratio of AUC(0-inf) after oral administration of ACT-541468 and after intravenous infusion of 14C-labeled ACT-541468 (tracer)

OTHER OUTCOMES:
Change from baseline in saccadic peak velocity (SPV) | At baseline till 10 hours after study drug administration
Change from baseline in body sway | At baseline till 10 hours after study drug administration
Change from baseline in adaptive tracking | At baseline till 10 hours after study drug administration
Chnage from baseline in Bond and Lader visual analog scale (B&L VAS)l | At baseline till 10 hours after study drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Clemens Muehlan, Study Director — Actelion
Locations (1):
- Investigator Site, Leiden, Netherlands